CLINICAL TRIAL: NCT02863419
Title: Efficacy and Safety of Oral Semaglutide Versus Liraglutide and Versus Placebo in Subjects With Type 2 Diabetes Mellitus
Acronym: PIONEER 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-4224; 2015-005210-30 (EudraCT Number); U1111-1176-6029 (Other: WHO)
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Results first posted 2019-11-07 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oral Semaglutide (Experimental)
  Interventions: Drug: semaglutide
- Liraglutide (Active Comparator)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Oral semaglutide once-daily.
  Arms: Oral Semaglutide
Drug: liraglutide — Subcutaneous (s.c.) injection once-daily.
  Arms: Liraglutide
Drug: placebo — Placebo once-daily.
  Arms: Placebo

SUMMARY:
This trial is conducted globally. The aim of this trial is to investigate efficacy and safety of oral Semaglutide versus Liraglutide and versus Placebo in Subjects with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, age above or equal to 18 years at the time of signing informed consent. For Japan only: Male or female, age at least 20 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus for at least 90 days prior to day of screening.
* HbA1c (glycosylated haemoglobin) of 7.0-9.5 % (53-80.3 mmol/mol) (both inclusive)
* Stable daily dose of metformin (above or equal to 1500 mg or maximum tolerated dose as documented in the subject medical record) alone or in combination with a stable daily dose of a SGLT-2 (sodium-glucose co-transporter-2) inhibitor for at least 90 days prior to day of screening (fixed-dose combinations are allowed)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice).For certain specific countries: Additional specific requirements apply
* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Family or personal history of Multiple Endocrine Neoplasia Type 2 (MEN 2) or Medullary Thyroid Carcinoma (MTC)
* History of pancreatitis (acute or chronic)
* History of major surgical procedures involving the stomach and potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* Any of the following: myocardial infarction (MI), stroke or hospitalisation for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Subjects with ALT (alanine aminotransferase) above 2.5 × upper normal limit (UNL)
* Renal impairment defined as estimated Glomerular Filtration Rate (eGFR) below 60 mL/min/1.73 m^2 as per Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI)
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before the day of screening. An exception is short-term insulin treatment for acute illness for a total of below or equal to 14 days
* Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or dilated fundoscopy performed within 90 days prior to randomisation
* History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and carcinoma in situ)
* History of diabetic ketoacidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-08-19 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (100):
- United States (37):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Los Alamitos, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Hallandale, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Ormond Beach, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Lebanon, New Hampshire
  - Novo Nordisk Investigational Site, Teaneck, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Mineola, New York
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Morganton, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Dublin, Ohio
  - Novo Nordisk Investigational Site, Maumee, Ohio
  - Novo Nordisk Investigational Site, Norman, Oklahoma
  - Novo Nordisk Investigational Site, McMurray, Pennsylvania
  - Novo Nordisk Investigational Site, Summerville, South Carolina
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, North Richland Hills, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Virginia Beach, Virginia
- Croatia (4):
  - Novo Nordisk Investigational Site, Karlovac
  - Novo Nordisk Investigational Site, Osijek
  - Novo Nordisk Investigational Site, Slavonski Brod
  - Novo Nordisk Investigational Site, Zagreb
- Czechia (3):
  - Novo Nordisk Investigational Site, Náchod
  - Novo Nordisk Investigational Site, Pilsen
  - Novo Nordisk Investigational Site, Prague
- Germany (8):
  - Novo Nordisk Investigational Site, Bochum
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Oldenburg I. Holst
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Villingen-Schwenningen
- Hungary (9):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Gyula
  - Novo Nordisk Investigational Site, Kalocsa
  - Novo Nordisk Investigational Site, Nagykanizsa
  - Novo Nordisk Investigational Site, Szeged
  - Novo Nordisk Investigational Site, Székesfehérvár
  - Novo Nordisk Investigational Site, Szigetvár
  - Novo Nordisk Investigational Site, Szolnok
  - Novo Nordisk Investigational Site, Tatabánya
- Japan (9):
  - Novo Nordisk Investigational Site, Bunkyo-ku, Tokyo
  - Novo Nordisk Investigational Site, Kumamoto-shi,Kumamoto
  - Novo Nordisk Investigational Site, Mito-shi, Ibaraki
  - Novo Nordisk Investigational Site, Okawa-shi, Fukuoka
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Tochigi
  - Novo Nordisk Investigational Site, Yamato-shi, Kanagawa
- Latvia (2):
  - Novo Nordisk Investigational Site, Ogre
  - Novo Nordisk Investigational Site, Riga
- Poland (9):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Bydgoszcz
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Gniewkowo
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Novo Nordisk Investigational Site, Toa Baja, Puerto Rico
- Slovakia (6):
  - Novo Nordisk Investigational Site, Bardejov
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Nitra
  - Novo Nordisk Investigational Site, Rožňava
  - Novo Nordisk Investigational Site, Vrútky
- South Africa (4):
  - Novo Nordisk Investigational Site, Benoni, Gauteng
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- Ukraine (3):
  - Novo Nordisk Investigational Site, Kyiv
  - Novo Nordisk Investigational Site, Odesa
  - Novo Nordisk Investigational Site, Vinnytsia
- United Arab Emirates (5):
  - Novo Nordisk Investigational Site, Ajman
  - Novo Nordisk Investigational Site, Al Mafraq
  - Novo Nordisk Investigational Site, Dubai
  - Novo Nordisk Investigational Site, Rahba City
  - Novo Nordisk Investigational Site, Umm Al Quwain City

REFERENCES:
- [Result] Pratley R, Amod A, Hoff ST, Kadowaki T, Lingvay I, Nauck M, Pedersen KB, Saugstrup T, Meier JJ; PIONEER 4 investigators. Oral semaglutide versus subcutaneous liraglutide and placebo in type 2 diabetes (PIONEER 4): a randomised, double-blind, phase 3a trial. Lancet. 2019 Jul 6;394(10192):39-50. doi: 10.1016/S0140-6736(19)31271-1. Epub 2019 Jun 8. PMID 31186120
- [Result] Araki E, Terauchi Y, Watada H, Deenadayalan S, Christiansen E, Horio H, Kadowaki T. Efficacy and safety of oral semaglutide in Japanese patients with type 2 diabetes: A post hoc subgroup analysis of the PIONEER 1, 3, 4 and 8 trials. Diabetes Obes Metab. 2021 Dec;23(12):2785-2794. doi: 10.1111/dom.14536. Epub 2021 Sep 27. PMID 34472698
- [Result] Aroda VR, Bauer R, Christiansen E, Haluzik M, Kallenbach K, Montanya E, Rosenstock J, Meier JJ. Efficacy and safety of oral semaglutide by subgroups of patient characteristics in the PIONEER phase 3 programme. Diabetes Obes Metab. 2022 Jul;24(7):1338-1350. doi: 10.1111/dom.14710. Epub 2022 May 9. PMID 35373893
- [Derived] Ren H, Berry S, Malkin SJP, Hunt B, Bain S. Early use of oral semaglutide in the UK: A cost-effectiveness analysis versus continuing metformin and SGLT-2 inhibitor therapy. BMJ Open. 2023 Sep 29;13(9):e070473. doi: 10.1136/bmjopen-2022-070473. PMID 37775297
- [Derived] Pratley RE, Crowley MJ, Gislum M, Hertz CL, Jensen TB, Khunti K, Mosenzon O, Buse JB. Oral Semaglutide Reduces HbA1c and Body Weight in Patients with Type 2 Diabetes Regardless of Background Glucose-Lowering Medication: PIONEER Subgroup Analyses. Diabetes Ther. 2021 Apr;12(4):1099-1116. doi: 10.1007/s13300-020-00994-9. Epub 2021 Mar 4. PMID 33660198
- [Derived] Thethi TK, Pratley R, Meier JJ. Efficacy, safety and cardiovascular outcomes of once-daily oral semaglutide in patients with type 2 diabetes: The PIONEER programme. Diabetes Obes Metab. 2020 Aug;22(8):1263-1277. doi: 10.1111/dom.14054. Epub 2020 May 13. PMID 32267058
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 101 sites in 12 countries as follows:Croatia (5), Czech Republic (3), Germany (8), Hungary (9), Japan (9), Latvia (4), Poland (9), Slovakia (5), South Africa (5), Ukraine (3), United Arab Emirates (2), United States (39).
Pre-assignment Details: Data presented in "participant flow" is based on the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Groups:
- Oral Semaglutide 14 mg: Participants were to take once-daily oral semaglutide tablets for 52 weeks. Participants started oral semaglutide at 3 mg and were dose-escalated in 4-week increments until the final maintenance dose of 14 mg once-daily was reached (i.e. 3 mg from week 0 to week 4, 7 mg from week 4 to week 8 and 14 mg from week 8 to week 52). In addition, participants were to take liraglutide placebo once-daily as a subcutaneous injection (under the skin) from week 0 to week 52. Participants were to continue their anti-diabetic background medication (metformin alone or in combination with a sodium-glucose co-transporter-2 [SGLT-2] inhibitor) throughout the entire trial.
- Liraglutide 1.8 mg: Participants were to take once-daily liraglutide subcutaneous injection (under the skin) for 52 weeks. Participants started liraglutide at 0.6 mg and were dose-escalated in one-week increments until the final maintenance dose of 1.8 mg once-daily was reached (i.e. 0.6 mg from week 0 to week 1, 1.2 mg from week 1 to week 2 and 1.8 mg from week 2 to week 52). In addition, participants were to take oral semaglutide placebo tablets once-daily from week 0 to week 52. Participants were to continue their anti-diabetic background medication (metformin alone or in combination with a sodium-glucose co-transporter-2 [SGLT-2] inhibitor) throughout the entire trial.
- Placebo: Participants were to take both oral semaglutide placebo tablets and liraglutide placebo once-daily as a subcutaneous injection (under the skin) from week 0 to week 52. Participants were to continue their anti-diabetic background medication (metformin alone or in combination with a sodium-glucose co-transporter-2 [SGLT-2] inhibitor) throughout the entire trial.
Period: Overall Study
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Started | 285 | 284 | 142
Full Analysis Set (FAS) | 285 | 284 | 142
Safety Analysis Set (SAS) | 285 | 284 | 142
Completed | 277 | 274 | 134
Not Completed | 8 | 10 | 8
Not completed — Lost to Follow-up | 0 | 1 | 4
Not completed — Withdrawal by Subject | 5 | 5 | 3
Not completed — Died | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo | Total
Number analyzed (Participants) | 285 | 284 | 142 | 711
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56 (10) | 56 (10) | 57 (10) | 56 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 135 | 68 | 341
  Male | 147 | 149 | 74 | 370
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 18 | 5 | 40
  Not Hispanic or Latino | 268 | 266 | 137 | 671
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race was recorded as 'Not Applicable' for South Africa.
  Participants
    White | 208 | 212 | 99 | 519
    Black or African American | 12 | 9 | 8 | 29
    Asian | 39 | 36 | 19 | 94
    American Indian or Alaska Native | 0 | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
    Other | 3 | 8 | 3 | 14
    Not Applicable | 23 | 17 | 12 | 52
Baseline HbA1c [Mean (Standard Deviation); unit: Percentage of HbA1c] — Observed mean HbA1c
  Percentage of HbA1c | 8.0 (0.7) | 8.0 (0.7) | 7.9 (0.7) | 8.0 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Week 26)
Description: Change from baseline (week 0) in glycosylated haemoglobin (HbA1c) was evaluated at week 26. The endpoint was evaluated based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. The endpoint was also evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Percentage of HbA1c
  In-trial: number analyzed (Participants) | 278 | 272 | 134
  In-trial | -1.2 (0.9) | -1.1 (0.9) | -0.1 (0.7)
  On-treatment without rescue medication: number analyzed (Participants) | 238 | 245 | 112
  On-treatment without rescue medication | -1.4 (0.9) | -1.2 (0.9) | -0.1 (0.7)
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Liraglutide 1.8 mg; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an analysis of covariance (ANCOVA) model with treatment, strata, and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Non-Inferiority — This hypothesis was controlled for multiplicity. Results are based on the data from the in-trial observation period. The estimated treatment effect includes the effect of any rescue medication and any effect after premature trial product discontinuation (treatment policy estimand). A value of 0.4% (the non-inferiority margin) was added to imputed values at week 26 for the oral semaglutide treatment arm only; p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from the non-inferiority margin. The non-inferiority margin was 0.4%; Mean treatment difference = -0.1, 95% CI 2-sided [-0.3 to 0.0] — Oral semaglutide 14 mg - Liraglutide 1.8 mg
Statistical Analysis 2: Comparison: Oral Semaglutide 14 mg vs Liraglutide 1.8 mg; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an ANCOVA model with treatment, strata, and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — This hypothesis was controlled for multiplicity. Results are based on the data from the in-trial observation period. The estimated treatment effect includes the effect of any rescue medication and any effect after premature trial product discontinuation (treatment policy estimand); p = 0.0645, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -0.1, 95% CI 2-sided [-0.3 to 0.0] — Oral semaglutide 14 mg - Liraglutide 1.8 mg
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -1.1, 95% CI 2-sided [-1.2 to -0.9] — Oral semaglutide 14 mg - Placebo
Statistical Analysis 4: Comparison: Oral Semaglutide 14 mg vs Liraglutide 1.8 mg; The analysis was based on a mixed model for repeated measurements (MMRM) that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment, strata and region as categorical fixed effects and the baseline HbA1c value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Non-Inferiority — This hypothesis was not controlled for multiplicity. Results are based on the data from the on-treatment without rescue medication observation period. The estimated treatment effect excludes the effect of any rescue medication and any effect after premature trial product discontinuation (hypothetical estimand); p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from the non-inferiority margin (non-inferiority). The non-inferiority margin was 0.4%; Mean treatment difference = -0.2, 95% CI 2-sided [-0.3 to -0.1] — Oral semaglutide 14 mg - Liraglutide 1.8 mg
Statistical Analysis 5: Comparison: Oral Semaglutide 14 mg vs Liraglutide 1.8 mg; [analysis description as in outcome 1, analysis 4]; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.0056, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -0.2, 95% CI 2-sided [-0.3 to -0.1] — Oral semaglutide 14 mg - Liraglutide 1.8 mg
Statistical Analysis 6: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -1.2, 95% CI 2-sided [-1.4 to -1.0] — Oral semaglutide 14 mg - Placebo

2. Secondary Outcome: Change in Body Weight (Week 26)
Description: Change from baseline (week 0) in body weight was evaluated at week 26. The endpoint was evaluated based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. The endpoint was also evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = FAS which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Kg
  In-trial: number analyzed (Participants) | 278 | 271 | 134
  In-trial | -4.4 (4.4) | -3.2 (3.7) | -0.6 (3.1)
  On-treatment without rescue medication: number analyzed (Participants) | 238 | 244 | 112
  On-treatment without rescue medication | -4.7 (4.3) | -3.3 (3.7) | -0.7 (3.1)
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Liraglutide 1.8 mg; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an ANCOVA model with treatment, strata, and region as categorical fixed effects and baseline body weight value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.0003, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -1.2, 95% CI 2-sided [-1.9 to -0.6] — Oral semaglutide 14 mg - Liraglutide 1.8 mg
Statistical Analysis 2: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -3.8, 95% CI 2-sided [-4.7 to -3.0] — Oral semaglutide 14 mg - Placebo
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Liraglutide 1.8 mg; The analysis was based on a MMRM that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment, strata and region as categorical fixed effects and the baseline body weight value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -1.5, 95% CI 2-sided [-2.2 to -0.9] — Oral semaglutide 14 mg - Liraglutide 1.8 mg
Statistical Analysis 4: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -4.0, 95% CI 2-sided [-4.8 to -3.2] — Oral sema 14 mg - Placebo

3. Secondary Outcome: Change in HbA1c (Week 52)
Description: Change from baseline (week 0) in HbA1c was evaluated at 52 weeks. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 275 | 269 | 133
Percentage of HbA1c | -1.2 (1.0) | -0.9 (1.0) | -0.1 (0.9)

4. Secondary Outcome: Change in Body Weight (Week 52)
Description: Change from baseline (week 0) in body weight was evaluated at 52 weeks. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 275 | 269 | 133
Kg | -4.4 (5.5) | -3.1 (4.4) | -1.0 (3.8)

5. Secondary Outcome: Change in Body Weight (%)
Description: Relative change from baseline (week 0) in body weight (kg) was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, Week 26, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Percentage change
  Week 26: number analyzed (Participants) | 278 | 271 | 134
  Week 26 | -4.89 (4.95) | -3.33 (3.78) | -0.60 (3.34)
  Week 52: number analyzed (Participants) | 275 | 269 | 133
  Week 52 | -4.94 (6.37) | -3.25 (4.33) | -0.99 (4.12)

6. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change from baseline (week 0) in fasting plasma glucose (FPG) was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
mmol/L
  Week 26: number analyzed (Participants) | 276 | 269 | 133
  Week 26 | -2.04 (2.28) | -1.91 (2.05) | -0.33 (2.03)
  Week 52: number analyzed (Participants) | 273 | 269 | 132
  Week 52 | -1.91 (2.41) | -1.54 (2.41) | -0.66 (1.99)

7. Secondary Outcome: Change in Body Mass Index
Description: Change from baseline (week 0) in body mass index (BMI) was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
kg/m^2
  Week 26: number analyzed (Participants) | 278 | 271 | 134
  Week 26 | -1.6 (1.6) | -1.1 (1.3) | -0.2 (1.1)
  Week 52: number analyzed (Participants) | 275 | 269 | 133
  Week 52 | -1.6 (2.0) | -1.1 (1.5) | -0.4 (1.4)

8. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
cm
  Week 26: number analyzed (Participants) | 278 | 269 | 134
  Week 26 | -4.2 (5.4) | -3.0 (4.5) | -1.2 (3.9)
  Week 52: number analyzed (Participants) | 275 | 266 | 133
  Week 52 | -4.4 (6.1) | -2.7 (5.1) | -1.7 (4.7)

9. Secondary Outcome: Change in Total Cholesterol - Ratio to Baseline
Description: Change from baseline (week 0) in total cholesterol (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Ratio of total cholesterol
  Week 26: number analyzed (Participants) | 277 | 267 | 134
  Week 26 | 0.96 (20.3) | 0.97 (21.6) | 0.99 (17.0)
  Week 52: number analyzed (Participants) | 274 | 264 | 133
  Week 52 | 0.98 (20.5) | 0.98 (19.6) | 1.02 (18.3)

10. Secondary Outcome: Change in Low-density Lipoprotein (LDL) Cholesterol - Ratio to Baseline
Description: Change from baseline (week 0) in low-density lipoprotein (LDL) cholesterol (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Ratio of LDL cholesterol
  Week 26: number analyzed (Participants) | 277 | 267 | 133
  Week 26 | 0.95 (29.9) | 0.97 (43.6) | 0.99 (30.8)
  Week 52: number analyzed (Participants) | 274 | 264 | 132
  Week 52 | 0.99 (31.6) | 1.00 (38.5) | 1.06 (33.1)

11. Secondary Outcome: Change in Very Low Density Lipoprotein (VLDL) Cholesterol - Ratio to Baseline
Description: Change from baseline (week 0) in VLDL cholesterol (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Ratio of VLDL cholesterol
  Week 26: number analyzed (Participants) | 277 | 267 | 133
  Week 26 | 0.90 (43.5) | 0.91 (37.1) | 1.02 (29.4)
  Week 52: number analyzed (Participants) | 274 | 264 | 132
  Week 52 | 0.87 (41.9) | 0.90 (37.5) | 0.98 (39.8)

12. Secondary Outcome: Change in High-density Lipoprotein (HDL) Cholesterol - Ratio to Baseline
Description: Change from baseline (week 0) in HDL cholesterol (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL-cholesterol
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Ratio of HDL-cholesterol
  Week 26: number analyzed (Participants) | 277 | 267 | 134
  Week 26 | 1.02 (13.8) | 1.02 (15.2) | 1.02 (12.2)
  Week 52: number analyzed (Participants) | 274 | 264 | 133
  Week 52 | 1.03 (13.8) | 1.01 (14.7) | 1.00 (12.7)

13. Secondary Outcome: Change in Triglycerides - Ratio to Baseline
Description: Change from baseline (week 0) in triglycerides (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Ratio of triglycerides
  Week 26: number analyzed (Participants) | 277 | 267 | 134
  Week 26 | 0.89 (48.4) | 0.91 (38.3) | 1.01 (34.7)
  Week 52: number analyzed (Participants) | 274 | 264 | 133
  Week 52 | 0.87 (47.0) | 0.89 (41.1) | 0.97 (43.4)

14. Secondary Outcome: Change in Free Fatty Acids - Ratio to Baseline
Description: Change from baseline (week 0) in free fatty acids (FFA) (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of FFA
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Ratio of FFA
  Week 26: number analyzed (Participants) | 271 | 262 | 132
  Week 26 | 0.94 (48.0) | 0.95 (50.7) | 1.06 (49.1)
  Week 52: number analyzed (Participants) | 270 | 261 | 130
  Week 52 | 0.83 (49.3) | 0.87 (51.2) | 0.89 (46.8)

15. Secondary Outcome: Change in SMPG - Mean 7-point Profile
Description: Change from baseline (week 0) to week 26 and week 52 in mean 7-point self-measured plasma glucose (SMPG) profile. SMPG was recorded at the following 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after dinner and at bedtime. Mean 7-point profile was defined as the area under the profile, calculated using the trapezoidal method, divided by the measurement time. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
mmol/L
  Week 26: number analyzed (Participants) | 263 | 257 | 129
  Week 26 | -2.2 (2.3) | -2.0 (2.0) | -0.7 (1.8)
  Week 52: number analyzed (Participants) | 263 | 251 | 126
  Week 52 | -2.2 (2.3) | -1.8 (2.2) | -0.9 (1.7)

16. Secondary Outcome: Change in SMPG - Mean Postprandial Increment Over All Meals
Description: Change from baseline (week 0) in the average of the post-prandial increments over all meals was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
mmol/L
  Week 26: number analyzed (Participants) | 264 | 257 | 129
  Week 26 | -0.7 (1.9) | -0.4 (2.0) | -0.2 (1.9)
  Week 52: number analyzed (Participants) | 264 | 253 | 126
  Week 52 | -0.5 (1.9) | -0.5 (2.1) | -0.4 (1.9)

17. Secondary Outcome: Participants Who Achieve HbA1c <7.0% (53 mmol/Mol) ADA Target (Yes/no)
Description: Participants who achieved HbA1c <7.0% (American Diabetes Association (ADA) target) (yes/no), was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Participants
  Week 26: number analyzed (Participants) | 278 | 272 | 134
  Week 26: Yes | 188 | 168 | 19
  Week 26: No | 90 | 104 | 115
  Week 52: number analyzed (Participants) | 275 | 269 | 133
  Week 52: Yes | 167 | 148 | 20
  Week 52: No | 108 | 121 | 113

18. Secondary Outcome: Participants Who Achieve HbA1c <6.5% (48 mmol/Mol) AACE Target (Yes/no)
Description: Participants who achieved HbA1c less than or equal to 6.5% (American Association of Clinical Endocrinologists (AACE) target) (yes/no) at weeks 26 and 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Participants
  Week 26: number analyzed (Participants) | 278 | 272 | 134
  Week 26: Yes | 133 | 116 | 7
  Week 26: No | 145 | 156 | 127
  Week 52: number analyzed (Participants) | 275 | 269 | 133
  Week 52: Yes | 119 | 88 | 5
  Week 52: No | 156 | 181 | 128

19. Secondary Outcome: Participants Who Achieve Weight Loss ≥5% (Yes/no)
Description: Participants who achieved weight loss more than or equal to 5% of their baseline body weight (yes/no) at weeks 26 and 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Participants
  Week 26: number analyzed (Participants) | 278 | 271 | 134
  Week 26: Yes | 121 | 75 | 10
  Week 26: No | 157 | 196 | 124
  Week 52: number analyzed (Participants) | 275 | 269 | 133
  Week 52: Yes | 123 | 66 | 16
  Week 52: No | 152 | 203 | 117

20. Secondary Outcome: Participants Who Achieve Weight Loss ≥ 10% (Yes/no)
Description: Participants who achieved weight loss more than or equal to 10% of their baseline body weight (yes/no) at weeks 26 and 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Participants
  Week 26: number analyzed (Participants) | 278 | 271 | 134
  Week 26: Yes | 39 | 16 | 0
  Week 26: No | 239 | 255 | 134
  Week 52: number analyzed (Participants) | 275 | 269 | 133
  Week 52: Yes | 45 | 20 | 4
  Week 52: No | 230 | 249 | 129

21. Secondary Outcome: Participants Who Achieve HbA1c <7.0 % (53 mmol/Mol) Without Hypoglycaemia (Severe or BG Confirmed Symptomatic Hypoglycaemia) and no Weight Gain (Yes/no)
Description: Participants who achieved HbA1c less than 7.0 % without severe or blood glucose (BG) confirmed symptomatic hypoglycaemia and without weight gain (yes/no) at weeks 26 and 52 are presented. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia was defined as an episode with plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Participants
  Week 26: number analyzed (Participants) | 278 | 271 | 134
  Week 26: Yes | 169 | 145 | 15
  Week 26: No | 109 | 126 | 119
  Week 52: number analyzed (Participants) | 275 | 269 | 133
  Week 52: Yes | 155 | 130 | 15
  Week 52: No | 120 | 139 | 118

22. Secondary Outcome: Participants Who Achieve HbA1c Reduction ≥1% (10.9 mmol/Mol) and Weight Loss ≥3% (Yes/no)
Description: Participants who achieved HbA1c reduction more than or equal to 1% of their baseline HbA1c and weight loss of more than or equal to 3% of their baseline body weight (yes/no) at weeks 26 and 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Participants
  Week 26: number analyzed (Participants) | 278 | 271 | 134
  Week 26: Yes | 130 | 93 | 5
  Week 26: No | 148 | 178 | 129
  Week 52: number analyzed (Participants) | 275 | 269 | 133
  Week 52: Yes | 120 | 77 | 9
  Week 52: No | 155 | 192 | 124

23. Secondary Outcome: Time to Additional Anti-diabetic Medication
Description: Presented results are the number of participants who had taken additional anti-diabetic medication anytime during the periods, from week 0 to week 26 and week 0 to week 52. Additional anti-diabetic medication was defined as any new anti-diabetic medication used for more than 21 days with the initiation at or after randomisation (week 0) and before (planned) end-of-treatment (week 52), and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before (planned) end-of-treatment. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Participants
  Week 0 to week 26 | 20 | 16 | 12
  Week 0 to week 52 | 39 | 29 | 46
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Liraglutide 1.8 mg; Time to initiation of additional anti-diabetic medication was analysed using a Cox proportional hazards model with treatment, strata, and region as categorical fixed effects and baseline HbA1c as covariate. Withdrawal for any reason or lost to follow-up contributed to the analysis as events (initiation of additional anti-diabetic medication). Censoring time was one day before planned end of treatment; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.4915, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.75 to 1.80] — Oral semaglutide 14 mg / Liraglutide 1.8 mg
Statistical Analysis 2: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 23, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.21 to 0.48] — Oral semaglutide 14 mg / Placebo

24. Secondary Outcome: Time to Rescue Medication
Description: Presented results are the number of participants who had taken rescue medication anytime during the periods, from week 0 to week 26 and week 0 to week 52. Rescue medication was defined as any new anti-diabetic medication used as add-on to trial product and used for more than 21 days with the initiation at or after randomisation (week 0) and before last day on trial product, and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before last day on trial product. Results are based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Weeks 0-52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Participants
  Week 0 - week 26 | 10 | 9 | 11
  Week 0 - week 52 | 20 | 18 | 43
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Liraglutide 1.8 mg; Time to initiation of rescue medication was analysed using a Cox proportional hazards model with treatment, strata, and region as categorical fixed effects and baseline HbA1c as covariate. Censoring time was one day before last day on trial product; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.6252, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.62 to 2.22] — Oral semaglutide 14 mg / Liraglutide 1.8 mg
Statistical Analysis 2: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 24, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.15, 95% CI 2-sided [0.09 to 0.26] — Oral semaglutide 14 mg / Placebo

25. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) During Exposure to Trial Product
Description: Treatment emergent adverse events (TEAEs) were recorded from week 0 to week 57 (52-week treatment period plus the 5-week follow-up period). Adverse events (AEs) with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period: Time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = safety analysis set (SAS) which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Events | 973 | 927 | 300

26. Secondary Outcome: Change in Amylase - Ratio to Baseline
Description: Change from baseline (week 0) in amylase (units/litre (U/L)) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product. Number Analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Ratio of amylase
  Week 26: number analyzed (Participants) | 248 | 252 | 128
  Week 26 | 1.13 (24.9) | 1.11 (26.1) | 0.99 (23.1)
  Week 52: number analyzed (Participants) | 240 | 241 | 123
  Week 52 | 1.14 (27.4) | 1.10 (26.1) | 0.98 (21.9)

27. Secondary Outcome: Change in Lipase - Ratio to Baseline
Description: Change from baseline (week 0) in lipase (U/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Ratio of lipase
  Week 26: number analyzed (Participants) | 248 | 252 | 128
  Week 26 | 1.33 (53.3) | 1.40 (58.8) | 0.99 (45.7)
  Week 52: number analyzed (Participants) | 240 | 241 | 123
  Week 52 | 1.28 (59.3) | 1.32 (51.5) | 0.96 (44.2)

28. Secondary Outcome: Change in Pulse Rate
Description: Change from baseline (week 0) in pulse rate was evaluated at weeks 26 and 52. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Beats/min
  Week 26: number analyzed (Participants) | 248 | 255 | 128
  Week 26 | 2 (9) | 3 (11) | 0 (9)
  Week 52: number analyzed (Participants) | 241 | 247 | 123
  Week 52 | 2 (9) | 3 (9) | 0 (9)

29. Secondary Outcome: Change in SBP and DBP
Description: Change from baseline (week 0) in systolic blood pressure (SBP) and diastolic blood pressure (DBP) was evaluated at weeks 26 and 52. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
mmHg
  SBP: 26 weeks: number analyzed (Participants) | 248 | 255 | 128
  SBP: 26 weeks | -4 (13) | -4 (13) | -2 (13)
  SBP: 52 weeks: number analyzed (Participants) | 241 | 247 | 123
  SBP: 52 weeks | -3 (14) | -3 (13) | -0 (13)
  DBP: 26 weeks | -1 (9) | -0 (9) | -1 (9)
  DBP: 52 weeks: number analyzed (Participants) | 241 | 247 | 123
  DBP: 52 weeks | -1 (8) | -1 (9) | 0 (9)

30. Secondary Outcome: Change in ECG Evaluation
Description: Change from baseline (week 0) in electrocardiogram (ECG) was evaluated at weeks 26 and week 52. Change from baseline results are presented as shift in findings (normal, abnormal and not clinically significant (NCS) and abnormal and clinically significant (CS)) from week 0 to week 26 and week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Participants
  Normal (week 0) to normal (week 26): number analyzed (Participants) | 139 | 143 | 73
  Normal (week 0) to normal (week 26) | 130 | 123 | 67
  Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 139 | 143 | 73
  Normal (week 0) to abnormal NCS (week 26) | 19 | 20 | 6
  Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 139 | 143 | 73
  Normal (week 0) to abnormal CS (week 26) | 0 | 0 | 0
  Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 96 | 102 | 52
  Abnormal NCS (week 0) to normal (week 26) | 15 | 27 | 19
  Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 96 | 102 | 52
  Abnormal NCS (week 0) to abnormal NCS (week 26) | 81 | 75 | 33
  Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 96 | 102 | 52
  Abnormal NCS (week 0) to abnormal CS (week 26) | 0 | 0 | 0
  Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 5 | 11 | 3
  Abnormal CS (week 0) to normal (week 26) | 0 | 2 | 2
  Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 5 | 11 | 3
  Abnormal CS (week 0) to abnormal NCS (week 26) | 2 | 2 | 1
  Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 5 | 11 | 3
  Abnormal CS (week 0) to abnormal CS (week 26) | 3 | 7 | 0
  Normal (week 0) to Normal (week 52): number analyzed (Participants) | 145 | 138 | 70
  Normal (week 0) to Normal (week 52) | 113 | 123 | 64
  Normal (week 0) to Abnormal NCS (week 52): number analyzed (Participants) | 145 | 138 | 70
  Normal (week 0) to Abnormal NCS (week 52) | 31 | 14 | 5
  Normal (week 0) to Abnormal CS (week 52): number analyzed (Participants) | 145 | 138 | 70
  Normal (week 0) to Abnormal CS (week 52) | 1 | 1 | 1
  Abnormal NCS (week 0) to Normal (week 52): number analyzed (Participants) | 92 | 99 | 51
  Abnormal NCS (week 0) to Normal (week 52) | 19 | 26 | 14
  Abnormal NCS (week 0) to Abnormal NCS (week 52): number analyzed (Participants) | 92 | 99 | 51
  Abnormal NCS (week 0) to Abnormal NCS (week 52) | 73 | 73 | 37
  Abnormal NCS (week 0) to Abnormal CS (week 52): number analyzed (Participants) | 92 | 99 | 51
  Abnormal NCS (week 0) to Abnormal CS (week 52) | 0 | 0 | 0
  Abnormal CS (week 0) to Normal (week 52): number analyzed (Participants) | 4 | 9 | 3
  Abnormal CS (week 0) to Normal (week 52) | 0 | 3 | 2
  Abnormal CS (week 0) to Abnormal NCS (week 52): number analyzed (Participants) | 4 | 9 | 3
  Abnormal CS (week 0) to Abnormal NCS (week 52) | 1 | 1 | 1
  Abnormal CS (week 0) to Abnormal CS (week 52): number analyzed (Participants) | 4 | 9 | 3
  Abnormal CS (week 0) to Abnormal CS (week 52) | 3 | 5 | 0

31. Secondary Outcome: Change in Physical Examination
Description: Participants with physical examination findings, normal, abnormal NCS and abnormal CS at baseline (weeks -2) and weeks 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. Results are presented for the following examinations: 1) Cardiovascular system; 2) Central and peripheral nervous system; 3) Gastrointestinal system, incl. mouth; 4) General appearance; 5) Head, ears, eyes, nose, throat, neck; 6) Lymph node palpation; 7) Musculoskeletal system; 8) Respiratory system; 9) Skin; 10) Thyroid gland.
Time Frame: Week -2, week 52
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Participants
  1) Cardiovascular system (Week -2): Normal | 260 | 249 | 128
  1) Cardiovascular system (Week -2): Abnormal NCS | 23 | 26 | 12
  1) Cardiovascular system (Week -2): Abnormal CS | 2 | 9 | 2
  1) Cardiovascular system (Week 52): number analyzed (Participants) | 275 | 269 | 133
  1) Cardiovascular system (Week 52): Normal | 255 | 236 | 118
  1) Cardiovascular system (Week 52): Abnormal NCS | 19 | 24 | 15
  1) Cardiovascular system (Week 52): Abnormal CS | 1 | 9 | 0
  2) Central and peripheral nervous system (Week -2): Normal | 258 | 254 | 123
  2) Central and peripheral nervous system (Week -2): Abnormal NCS | 16 | 16 | 13
  2) Central and peripheral nervous system (Week -2): Abnormal CS | 11 | 14 | 6
  2) Central and peripheral nervous system (Week 52): number analyzed (Participants) | 275 | 269 | 133
  2) Central and peripheral nervous system (Week 52): Normal | 247 | 239 | 115
  2) Central and peripheral nervous system (Week 52): Abnormal NCS | 20 | 20 | 11
  2) Central and peripheral nervous system (Week 52): Abnormal CS | 8 | 10 | 7
  3) Gastrointestinal system, incl. mouth (Week -2): Normal | 275 | 271 | 133
  3) Gastrointestinal system, incl. mouth (Week -2): Abnormal NCS | 10 | 13 | 9
  3) Gastrointestinal system, incl. mouth (Week -2): Abnormal CS | 0 | 0 | 0
  3) Gastrointestinal system, incl. mouth (Week 52): number analyzed (Participants) | 275 | 269 | 133
  3) Gastrointestinal system, incl. mouth (Week 52): Normal | 266 | 260 | 123
  3) Gastrointestinal system, incl. mouth (Week 52): Abnormal NCS | 9 | 9 | 10
  3) Gastrointestinal system, incl. mouth (Week 52): Abnormal CS | 0 | 0 | 0
  4) General appearance (Week -2): Normal | 203 | 212 | 109
  4) General appearance (Week -2): Abnormal NCS | 67 | 54 | 22
  4) General appearance (Week -2): Abnormal CS | 15 | 18 | 11
  4) General appearance (Week 52): number analyzed (Participants) | 275 | 269 | 133
  4) General appearance (Week 52): Normal | 208 | 204 | 105
  4) General appearance (Week 52): Abnormal NCS | 59 | 55 | 20
  4) General appearance (Week 52): Abnormal CS | 8 | 10 | 8
  5) Head, ears, eyes, nose, throat, neck (Week -2): Normal | 275 | 269 | 138
  5) Head, ears, eyes, nose, throat, neck (Week -2): Abnormal NCS | 9 | 13 | 3
  5) Head, ears, eyes, nose, throat, neck (Week -2): Abnormal CS | 1 | 2 | 1
  5) Head, ears, eyes, nose, throat, neck (Week 52): number analyzed (Participants) | 275 | 268 | 132
  5) Head, ears, eyes, nose, throat, neck (Week 52): Normal | 267 | 258 | 129
  5) Head, ears, eyes, nose, throat, neck (Week 52): Abnormal NCS | 8 | 10 | 3
  5) Head, ears, eyes, nose, throat, neck (Week 52): Abnormal CS | 0 | 0 | 0
  6) Lymph node palpation (Week -2): Normal | 285 | 283 | 142
  6) Lymph node palpation (Week -2): Abnormal NCS | 0 | 1 | 0
  6) Lymph node palpation (Week -2): Abnormal CS | 0 | 0 | 0
  6) Lymph node palpation (Week 52): number analyzed (Participants) | 275 | 269 | 133
  6) Lymph node palpation (Week 52): Normal | 275 | 268 | 133
  6) Lymph node palpation (Week 52): Abnormal NCS | 0 | 1 | 0
  6) Lymph node palpation (Week 52): Abnormal CS | 0 | 0 | 0
  7) Musculoskeletal system (Week -2): Normal | 268 | 264 | 131
  7) Musculoskeletal system (Week -2): Abnormal NCS | 14 | 17 | 10
  7) Musculoskeletal system (Week -2): Abnormal CS | 3 | 3 | 1
  7) Musculoskeletal system (Week 52): number analyzed (Participants) | 275 | 268 | 132
  7) Musculoskeletal system (Week 52): Normal | 262 | 257 | 124
  7) Musculoskeletal system (Week 52): Abnormal NCS | 11 | 10 | 7
  7) Musculoskeletal system (Week 52): Abnormal CS | 2 | 1 | 1
  8) Respiratory system (Week -2): Normal | 282 | 278 | 140
  8) Respiratory system (Week -2): Abnormal NCS | 3 | 5 | 0
  8) Respiratory system (Week -2): Abnormal CS | 0 | 1 | 2
  8) Respiratory system (Week 52): number analyzed (Participants) | 275 | 269 | 133
  8) Respiratory system (Week 52): Normal | 273 | 262 | 131
  8) Respiratory system (Week 52): Abnormal NCS | 2 | 6 | 0
  8) Respiratory system (Week 52): Abnormal CS | 0 | 1 | 2
  9) Skin (Week -2): Normal | 243 | 243 | 122
  9) Skin (Week -2): Abnormal NCS | 40 | 36 | 17
  9) Skin (Week -2): Abnormal CS | 2 | 5 | 3
  9) Skin (Week 52): number analyzed (Participants) | 275 | 269 | 133
  9) Skin (Week 52): Normal | 243 | 235 | 114
  9) Skin (Week 52): Abnormal NCS | 30 | 30 | 17
  9) Skin (Week 52): Abnormal CS | 2 | 4 | 2
  10) Thyroid gland (Week -2): Normal | 276 | 277 | 132
  10) Thyroid gland (Week -2): Abnormal NCS | 5 | 5 | 8
  10) Thyroid gland (Week -2): Abnormal CS | 4 | 2 | 2
  10) Thyroid gland (Week 52): number analyzed (Participants) | 275 | 269 | 133
  10) Thyroid gland (Week 52): Normal | 267 | 262 | 127
  10) Thyroid gland (Week 52): Abnormal NCS | 5 | 6 | 4
  10) Thyroid gland (Week 52): Abnormal CS | 3 | 1 | 2

32. Secondary Outcome: Change in Eye Examination Category
Description: Participants with eye examination (fundoscopy) findings, normal, abnormal NCS and abnormal CS at baseline (week -2) and week 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week -2, Week 52
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Participants
  Left eye - Normal to Normal | 130 | 144 | 57
  Left eye - Normal to Abnormal NCS | 10 | 15 | 5
  Left eye - Normal to Abnormal CS | 4 | 4 | 2
  Left eye - Abnormal NCS to normal | 15 | 13 | 5
  Left eye - Abnormal NCS to abnormal NCS | 63 | 43 | 38
  Left eye - Abnormal NCS to abnormal CS | 1 | 1 | 1
  Left eye - Abnormal CS to normal | 1 | 3 | 0
  Left eye - Abnormal CS to abnormal NCS | 5 | 3 | 2
  Left eye - Abnormal CS to abnormal CS | 7 | 12 | 8
  Right eye - Normal to Normal | 127 | 150 | 57
  Right eye - Normal to Abnormal NCS | 10 | 13 | 7
  Right eye - Normal to Abnormal CS | 3 | 4 | 2
  Right eye - Abnormal NCS to Normal | 16 | 12 | 6
  Right eye - Abnormal NCS to Abnormal NCS | 64 | 42 | 37
  Right eye - Abnormal NCS to Abnormal CS | 2 | 1 | 1
  Right eye - Abnormal CS to Normal | 2 | 3 | 1
  Right eye - Abnormal CS to Abnormal NCS | 5 | 2 | 1
  Right eye - Abnormal CS to Abnormal CS | 7 | 11 | 6

33. Secondary Outcome: Occurrence of Anti-semaglutide Binding Antibodies (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Number of participants who measured with anti-semaglutide binding antibodies anytime during post-baseline visits (weeks 0-57) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 251
Participants | 0

34. Secondary Outcome: Occurrence of Anti-semaglutide Neutralising Antibodies (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Number of participants who measured with anti-semaglutide neutralising antibodies anytime during post-baseline visits (weeks 0-57) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 251
Participants | 0

35. Secondary Outcome: Occurrence of Anti-semaglutide Binding Antibodies Cross Reacting With Native GLP-1 (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Number of participants who measured with anti-semaglutide binding antibodies cross reacting with native glucagon-like peptide-1 (GLP-1) anytime during post-baseline visits (weeks 0-57) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0-57
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 251
Participants | 0

36. Secondary Outcome: Occurrence of Anti-semaglutide Neutralising Antibodies Cross Reacting With Native GLP-1 (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Number of participants who measured with anti-semaglutide neutralising antibodies cross reacting with native GLP-1 anytime during post-baseline visits (weeks 0-57) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 251
Participants | 0

37. Secondary Outcome: Anti-semaglutide Binding Antibody Levels
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. It is based on the data from participants who were measured with anti-semaglutide antibodies anytime during post-baseline visits (weeks 0-57). Results are presented as percentage of bound radioactivity-labelled semaglutide /total added radioactivity-labelled semaglutide (%B/T). Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-57
Population: Overall number of participants analysed = participants who were found positive for anti-semaglutide antibodies.
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 0

38. Secondary Outcome: Number of Treatment-emergent Severe or Blood Glucose-confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded during weeks 0-57 (52-week treatment period plus the 5-week follow-up period). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a subject was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Weeks 0-57
Population: as for outcome 32
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Episodes | 2 | 9 | 3

39. Secondary Outcome: Participants With Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded from week 0 to week 57 (52-week treatment period plus the 5-week follow-up period). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a subject was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Weeks 0-57
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Participants | 2 | 7 | 3

40. Secondary Outcome: Change in DTSQs: Individual Items and Total Treatment Satisfaction Score (6 of the 8 Items Summed)
Description: Change from baseline (week 0) in Diabetes Treatment Satisfaction Questionnaire - status version (DTSQs) was evaluated at week 26 (wk 26) and week 52 (wk 52). The DTSQs items are scored on a 7-point graded response scale ranging from 6 to 0. Higher scores indicate higher levels of treatment satisfaction for DTSQs items 1, 4 -8. For items 2 and 3 a higher score indicates a higher patient perceived experience of hyperglycaemia and hypoglycaemia, respectively. Thus, lower scores indicate a perception of blood glucose levels being "none of the time" unacceptably high (item 2) or low (item 3). The domain score of total treatment satisfaction (total treatment satisfaction score) was computed by adding the six items scores 1, 4-8. The score has a minimum of 0 and a maximum of 36. A higher treatment satisfaction score indicates a higher level of treatment satisfaction.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 285 | 284 | 142
Scores on a scale
  Satisfaction with treatment: wk 26: number analyzed (Participants) | 276 | 271 | 134
  Satisfaction with treatment: wk 26 | 0.72 (1.49) | 0.73 (1.54) | 0.28 (1.69)
  Satisfaction with treatment: wk 52: number analyzed (Participants) | 275 | 268 | 133
  Satisfaction with treatment: wk 52 | 0.67 (1.67) | 0.70 (1.46) | 0.48 (1.45)
  Feeling of unacceptably high blood sugars: wk 26: number analyzed (Participants) | 276 | 272 | 134
  Feeling of unacceptably high blood sugars: wk 26 | -1.94 (2.03) | -1.72 (2.10) | -0.87 (2.11)
  Feeling of unacceptably high blood sugars: wk 52: number analyzed (Participants) | 275 | 269 | 133
  Feeling of unacceptably high blood sugars: wk 52 | -1.97 (2.13) | -1.71 (2.11) | -1.04 (2.10)
  Feeling of unacceptably low blood sugars: wk 26: number analyzed (Participants) | 276 | 272 | 133
  Feeling of unacceptably low blood sugars: wk 26 | -0.18 (1.81) | 0.03 (1.90) | -0.07 (1.57)
  Feeling of unacceptably low blood sugars: wk 52: number analyzed (Participants) | 275 | 269 | 132
  Feeling of unacceptably low blood sugars: wk 52 | -0.17 (1.85) | -0.06 (1.75) | -0.14 (1.45)
  Convenience of treatment: wk 26: number analyzed (Participants) | 276 | 271 | 134
  Convenience of treatment: wk 26 | 0.55 (1.38) | 0.39 (1.48) | 0.17 (1.81)
  Convenience of treatment: wk 52: number analyzed (Participants) | 275 | 268 | 133
  Convenience of treatment: wk 52 | 0.50 (1.47) | 0.42 (1.44) | 0.21 (1.75)
  Flexibility of treatment: wk 26: number analyzed (Participants) | 276 | 271 | 134
  Flexibility of treatment: wk 26 | 0.45 (1.53) | 0.43 (1.48) | 0.09 (1.34)
  Flexibility of treatment: wk 52: number analyzed (Participants) | 275 | 268 | 133
  Flexibility of treatment: wk 52 | 0.38 (1.52) | 0.40 (1.62) | 0.14 (1.51)
  Satisfaction with understanding of diabetes: wk 26: number analyzed (Participants) | 276 | 272 | 134
  Satisfaction with understanding of diabetes: wk 26 | 0.66 (1.31) | 0.52 (1.37) | 0.38 (1.18)
  Satisfaction with understanding of diabetes: wk 52: number analyzed (Participants) | 275 | 269 | 133
  Satisfaction with understanding of diabetes: wk 52 | 0.65 (1.29) | 0.54 (1.41) | 0.27 (1.38)
  Recommending treatment to others: wk 26: number analyzed (Participants) | 276 | 271 | 134
  Recommending treatment to others: wk 26 | 0.57 (1.47) | 0.63 (1.59) | 0.10 (1.34)
  Recommending treatment to others: wk 52: number analyzed (Participants) | 275 | 268 | 133
  Recommending treatment to others: wk 52 | 0.60 (1.55) | 0.48 (1.61) | 0.02 (1.70)
  Satisfaction to continue present treatment: wk 26: number analyzed (Participants) | 276 | 271 | 134
  Satisfaction to continue present treatment: wk 26 | 0.64 (1.68) | 0.74 (1.76) | 0.22 (1.80)
  Satisfaction to continue present treatment: wk 52: number analyzed (Participants) | 275 | 268 | 133
  Satisfaction to continue present treatment: wk 52 | 0.60 (1.81) | 0.56 (1.74) | 0.11 (1.77)
  Total treatment satisfaction: wk 26: number analyzed (Participants) | 276 | 271 | 134
  Total treatment satisfaction: wk 26 | 3.59 (6.12) | 3.44 (6.51) | 1.24 (6.71)
  Total treatment satisfaction: wk 52: number analyzed (Participants) | 275 | 268 | 133
  Total treatment satisfaction: wk 52 | 3.41 (6.81) | 3.11 (6.93) | 1.23 (6.96)

ADVERSE EVENTS:
Time Frame: Week 0 to week 57 (52 weeks treatment period + 5 weeks follow-up period). Results are based on the safety analysis set (SAS), which comprised all randomised participants who received at least one dose of trial product.
Description: Serious adverse events and other AEs were based on the on-treatment observation period, i.e., the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. All-cause mortality were based on the in-trial observation period, i.e., the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Arm/Group | Oral Semaglutide 14 mg | Liraglutide 1.8 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 3/285 | 4/284 | 1/142
Serious Adverse Events (participants affected / at risk) | 31/285 | 22/284 | 15/142
Other Adverse Events (participants affected / at risk) | 148/285 | 120/284 | 47/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 14 mg (N=285) | Liraglutide 1.8 mg (N=284) | Placebo (N=142)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic haematoma (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Investigation (Investigations) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ligamentitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic vein thrombosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Oral fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 14 mg (N=285) | Liraglutide 1.8 mg (N=284) | Placebo (N=142)
Abdominal pain (Gastrointestinal disorders) | 16 (16) | 6 (6) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 17 (19) | 5 (6)
Blood glucose increased (Investigations) | 0 (0) | 2 (2) | 9 (10)
Constipation (Gastrointestinal disorders) | 22 (23) | 11 (12) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 16 (17) | 20 (23) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 43 (59) | 31 (42) | 11 (11)
Dyspepsia (Gastrointestinal disorders) | 16 (26) | 12 (13) | 0 (0)
Headache (Nervous system disorders) | 27 (33) | 17 (24) | 8 (12)
Nasopharyngitis (Infections and infestations) | 41 (60) | 37 (59) | 15 (18)
Nausea (Gastrointestinal disorders) | 55 (69) | 51 (67) | 5 (5)
Vomiting (Gastrointestinal disorders) | 24 (28) | 13 (24) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT02863419/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT02863419/SAP_001.pdf